CLINICAL TRIAL: NCT00040157
Title: A Phase 2 Trial of 4 Weeks of ACH-126,443 in Comparison With Continued Lamivudine in Stable Triple Antiretroviral Combination Therapy in HIV-Infected Subjects With Modestly Detectable Viral Load
Brief Title: Safety and Antiviral Study of ACH-126, 443 (Beta-L-Fd4C) in the Treatment of Adults With HIV Infection and Modestly Detectable Viral Load.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety concerns
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH443-006
Record Dates: First submitted 2002-06-21; First posted 2002-06-25 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infections
Keywords: treatment experienced,; Stable triple anti-retroviral combination therapy in HIV-infected,; Achillion
MeSH Terms: conditions — HIV Infections | interventions — dexelvucitabine

INTERVENTIONS:
Drug: ACH126-443 (Beta-L-Fd4C)

SUMMARY:
To determine safety and efficacy of ACH-126,443 on the treatment of adults with HIV infection who have modestly detectable viral load while on stable triple combination antiretroviral therapy including 3TC.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Receiving a stable triple combination antiretroviral regimen including 3TC, one other NRTI and either an NNRTI or a protease inhibitor for at least 4 months (16 weeks)
* Demonstration of initial viral suppression and subsequent rebound to be defined as an initial virological drop of at least 0.5 Logs on a 3TC-containing regimen
* Plasma HIV RNA level > 1000 and < 30,000 copies/mL on two occasions
* Genotypically documented M184V variant of HIV RT
* Clinically stable HIV status with no AIDS-defining events
* CD4 > 200 cells/mm3
* Basic hematologic and chemistry parameters within acceptable limits (defined in protocol)
* All women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L of b-HCG) within 72 hours prior to the start of study medication
* No active opportunistic infection requiring treatment
* Subject must be able to provide written informed consent
* Baseline laboratory values measured within 28 days of initiating study drug as follows:
* HGB≥9.0g/dl or HCT≥27% (in the absence of blood transfusions or erythropoietin treatment in the preceding two weeks
* Absolute neutrophil count≥1000 cells/mm(^3) (in the absence of on-going G-CSF therapy
* Platelet count ≥75,000/mm(^3)
* AST <7.0 times the upper limit of normal
* ALT ,7.0 times the upper limit of normal
* Serum creatinine <1.1 times the upper limit of normal

Exclusion Criteria

* Evidence of active HBV infection as demonstrated by HBsAg positivity
* Hepatitis C co-infection
* Concurrent systemic antiviral treatment
* Previous therapy with agents with significant systemic myelosuppressive or cytotoxic potential within 3 months of study start or the expected need for such therapy at study start.
* Alcohol abuse
* Pregnancy or breast-feeding
* Inability to tolerate oral medication
* AST > 7.0 times the upper limit of normal
* ALT > 7.0 times the upper limit of normal
* Any clinical condition or prior therapy that, in the Investigators opinion, would make the subject unsuitable for the study or unable to comply with the dosing requirements.
* Use of any other drug or substance with anti-HBV activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Body Positive, Inc., Phoenix, Arizona
  - Los Angeles, California
  - Pacific Horizon Medical Group, Inc., San Francisco, California
  - Community Health Care Center One, Inc., Fort Lauderdale, Florida
  - South Shore Hospital, Miami Beach, Florida
  - AIDS Research Consortium, Atlanta, Georgia
  - Chicago, Illinois
  - St. Lukes Roosevelt Hospital, New York, New York
  - Stony Brook University Infectious Disease, Dept. of Medicine, Stony Brook, New York
  - Houston, Texas
  - Hampton Road Medical Specialists, Hampton, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.achillion.com